CLINICAL TRIAL: NCT07352254
Title: OutreAch MediCal Care for HousEbound Patients With Post-COVID-19 Syndrome or ME/CFS of Any Cause
Brief Title: OutreAch MediCal Care for HousEbound Patients With Post-COVID-19 Syndrome or ME/CFS of Any Cause (ACCESS)
Acronym: ACCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Bundesministerium für Gesundheit, Familie und Jugend (Unknown)
Responsible Party: Principal Investigator, Dirks, Meike Dr., Consultant, Department of Neurology, Principal Investigator, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11793-BO-S-2025
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: ME/CFS
Keywords: ME/CFS; housebound; house call
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensified medical care (Experimental): monthly online visit in addition to standard care
  Interventions: Other: online visit
- standard care (Active Comparator): standard care as decided after discussion between family doctor and visiting specialists
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: online visit — monthly online visits
  Arms: intensified medical care
Other: No Interventions — No Interventions
  Arms: standard care

SUMMARY:
The significance of the Post-COVID Syndrome (PCS) has been widely acknowledged. Various efforts are made to find out about the pathomechanisms behind PCS and to establish therapies. One sub-group of PCS-patients, however, is generally excluded from any studies, and that are those who are unable to visit outpatient clinics or hospitals for diagnostic work up or participation in clinical trials, as they are unable to leave their home and to seek medical support on their own physical and mental capabilities. They are housebound, mostly or totally bedridden. Similar cases are known from myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) of any cause and are graded as moderate to very severe ME/CFS according to the Canadian Consensus criteria. The patients are usually seen by their family doctor and have no access to medical specialists.

The planned project aims to find out about the prevalence of this most severe manifestation of PCS, the clinical characteristics, the prevalence of mimics, risk factors and impact of the disease on the patients' life and their family/caregivers. Individual care and treatment plans will be developed and the effect of monthly consultation hours for patients and caregivers upon the patients' health status and the caregiver burden will be evaluated in a randomized controlled trial. The project will be performed in close cooperation between patients, caregivers, the patient's family doctor and a board of experts from internal medicine, neurology, psychosomatic medicine and general medicine at Hannover Medical School.

We expect an improvement of the patients' and caregivers wellbeing with intensified medical care. We are aware, however, that intensification of the patient-doctor interaction carries the risk to exacerbate the patients' symptoms. The results of our study will show how current models of care for PCS and ME/CFS patients should be modified to fit to the individual patient's aims and capacities.

DETAILED DESCRIPTION:
Based on own clinical experience the grant applicants notice a deficit in the current medical care for patients with Post-COVID Syndrome as well as patients with ME/CFS of other causes, who are unable to leave their home -some of them even bedridden - due to extreme fatigue and exhaustibility. Therefore, we developed a multi-disciplinary project focussed on the as-sessment of prevalence and special needs of this patient group, that - in case of a positive evaluation - can easily be transferred into routine medical care.

The planned project aims are:

1. to characterize the main clinical symptoms of the extreme PCS or ME/CFS variant

   * via standardized anamnesis and physical and mental assessment by specialists in internal medicine, neurology and psychosomatic medicine performed at separate home visits of the patients. In addition to the patients also the caregivers will be interviewed in standardized manner regarding symptom onset and development.
   * Patients will be recruited via their family doctors, patient support groups and social media as well as through our Post-COVID outpatient clinics through calls we get from housebound patients and their caretakers.
2. to detect and describe PCS/ME/CFS mimics in this group of patients

   * via the analysis of all data achieved from home visits as well as the available data of former diagnostic efforts in cooperation with the responsible family doctor.
   * Our structured care at Outreach Medical Care for ME/CFS patients includes a thorough evaluation of previous medical findings, where available. Findings that were made years before the onset of symptoms may also be relevant. These findings are recorded in a structured form and are included in the evaluation. Since the electronic health record shall be compiled for every member of a statutory health insurance until January 2025 previous medical findings should be more easily available than currently.
3. to identify possible risk factors for the development of the extreme PCS or ME/CFS variant

   - via the comparison of characteristics such as age, sex, BMI, accompanying diseases, the patients' medical history as well as socio-economic status including level of education, occupation, household income of the patients recruited into the planned study to already available data on subjects with a COVID-19 history but no (n=88) or less severe Post-COVID symptoms (n=115) evaluated at the Department of Neurology, recently.
4. to assess the impact of the moderate to very severe ME/CFS or PCS upon the patients' daily living activities (ADL) and their health-related quality of life (HRQoL)

   - via the self-report questionnaires Functional Independence Measure (FIM), a weighted activity score developed for ME/CFS patients for ADL and SF-36 for HRQoL.
5. to assess the caregiver burden associated with the patients' 24/7 need for support

   - via the Zarit Burden Interview
6. to develop individual care and treatment plans for every patient

   * via online discussion of every case in an interdisciplinary board consisting of the specialists in internal medicine, neurology and psychosomatic medicine, who have examined the pa-tients during the home visit, the patient's family doctor, and a team of specialists involved in the care for PCS patients at the PCS out-patient clinic at Hannover Medical School (a social worker, a general practitioner and specialists for pulmonology, rheumatology and rehabilita-tion medicine). This board shall act as a bridge between highly specialised university medi-cine and primary care.
   * Of note, patients will be included into the study only if their caregiver and their family doctor agree to take part as well.
7. to evaluate the effect of monthly consultation hours for patients and caregivers upon the patients' health status and the caregiver burden in a randomized controlled trial - The primary objective of the randomized controlled trial (RCT) is to compare extensive vs. non-extensive care of patients and caregivers. In the non-extensive group patients will be visited at baseline and will receive their individual treatment plan that is prescribed and mon-itored by their family doctor. In the extensive care group patients and caregivers will receive extensive support for the realization of the treatment plan by the ACCESS study team includ-ing the opportunity for online consultations held by one specialist of the three involved disci-plines every month. The effect of the extensive care shall be evaluated by self-report questionnaires of physical and mental health related quality of life (SF36), ADL and caregiver burden in both groups 3, 6, 9 and 12 months after randomization. Moreover, the patients' clinical status shall be assessed 1 year after randomization via rerun of the examinations performed at baseline during a home visit.

For the assessment of long-term effects a further online follow-up will be performed 24 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* ME/CFS according to the Canadian Consensus Criteria
* Bell Score ≤ 30
* Duration of the postexertional malaise (PEM) > 14 hours
* Age > 18 years and < 70

Exclusion Criteria:

- Pre-existing conditions or comorbidities that have (or could have) led to a restriction of mobility or mental capacity, such as various diseases of the central nervous system.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Short Form (SF)-36 health survey, physical score | 1 year
  Short-Form (SF-36) health survey to assess health related quality of life, here the physical score. Higher values indicate better health status. The range depends on age, gender and education.

CONTACTS AND LOCATIONS:
Overall Officials: Meike Dirks, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the data with the registry of the outpatient clinic for rare diseases at MHH
Supporting Information: Study Protocol, ICF
Time Frame: The IPD and supporting information will be available after final data analysis for ACCESS for at least 10 years
Access Criteria: Anonymous data will be available for scientific purposes after reasonable request

REFERENCES:
- [Result] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Result] Braun M, Scholz U, Hornung R, Martin M. The burden of spousal caregiving: a preliminary psychometric evaluation of the German version of the Zarit burden interview. Aging Ment Health. 2010 Mar;14(2):159-67. doi: 10.1080/13607860802459781. PMID 20336547
- [Result] Morfeld M, Kirchberger I, Bullinger M. SF-36- Fragebogen zum Gesundheitszustand, 2. Auflage, Hogrefe Verlag, 2011
- [Result] Buldyrev SV, Goldberger AL, Havlin S, Mantegna RN, Matsa ME, Peng CK, Simons M, Stanley HE. Long-range correlation properties of coding and noncoding DNA sequences: GenBank analysis. Phys Rev E Stat Phys Plasmas Fluids Relat Interdiscip Topics. 1995 May;51(5):5084-91. doi: 10.1103/physreve.51.5084. PMID 9963221
- [Result] Keith RA, Granger CV, Hamilton BB, Sherwin FS. The functional independence measure: a new tool for rehabilitation. Adv Clin Rehabil. 1987;1:6-18. No abstract available. PMID 3503663